CLINICAL TRIAL: NCT04109937
Title: A Phase III Multicenter Randomized Trial Assessing the Efficacy of Post-Operative Conventional External Beam Radiation Therapy Following Orthopaedic Surgery in Patients With Lower Extremity Bone Metastases
Brief Title: External Beam Radiation Therapy Post Surgery in Patients With Lower Extremity Bone Metastases Randomized Efficacy Trial
Acronym: EXPLORE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Feasibility couldn't be worked out
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXPLORE
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Bone Metastases; Lower Extremity Fracture; Pathological Fracture; Impending Fracture
MeSH Terms: conditions — Fractures, Spontaneous

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive 1 of the 2 treatment arms.
Masking Description: Study is not blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery Alone (No Intervention): Patients with lower extremity bone metastases will receive surgical fixation/reconstruction but will not receive any post-operative radiation therapy.
- Surgery and Post-Operative Radiation Therapy (Active Comparator): Patients with lower extremity bone metastases will receive surgical fixation/reconstruction and will receive any post-operative radiation therapy.
  Interventions: Radiation: External beam radiation therapy

INTERVENTIONS:
Radiation: External beam radiation therapy — The post-operative radiation will cover entire prosthesis/surgical fixation device and will consist of the dose fractionation of: 20 Gy in 5 fractions or 30 Gy in 10 fractions.
  Arms: Surgery and Post-Operative Radiation Therapy

SUMMARY:
The objective of the present study is to evaluate the effectiveness of post-operative radiation therapy in lower extremity bone metastases. This trial will compare the health outcomes of patients receiving radiation therapy after Orthopaedic surgery to patients who will not receive radiation therapy post-surgery. The primary objective of the study is to compare the need for a subsequent surgery at the same treatment site within 12 months of the initial surgery. Additionally, the need for radiation or re-irradiation, functional status, performance status, pain scores, radiologically detected local disease progression, and overall length of survival will be compared at clinical endpoints for the two study arms. It is hypothesized that those randomized to receive post-operative radiation therapy will less likely need a subsequent surgery within the 12 months after the primary surgical intervention. This may optimize the quality of life for this patient population.

DETAILED DESCRIPTION:
The incidence of bone metastases in advanced cancer patients is substantial, representing 70% of all metastatic sites. Approximately 5-10% of all patients with bone metastases develop pathological fractures. Surgical reconstruction can be helpful following fracture or prophylactically in cases of an impending fracture. In these cases, post-operative radiation is the current clinical practice in North America and many countries around the world. Post-operative radiation has the potential to support bone healing and prevent tumor progression while also decreasing the need for subsequent orthopaedic surgeries to the same site. A recent systematic review, however, challenged the evidence on its efficacy and adoption as standard of care in this patient population. As well, post-operative radiation requires additional visits to the radiation centre (associated with added costs and efforts for both the patients and the healthcare system). There is also a "pain flare" phenomenon, in which up to 40% of patients receiving radiation for palliative bone metastases experience pain within 1-5 days following radiation. The pain can last for 10 days and may acutely mask potential clinical benefits of radiation.

Given that there is potential negative impact to these patients who are palliative with a relatively short lifespan, it is important that the efficacy of post-operative radiation is rigorously evaluated.

We propose a multicenter randomized controlled trial to assess the efficacy of post-operative radiation following orthopaedic surgery in patients with lower extremity bone metastases. 300 patients with pending or established lower extremity pathological fracture will be recruited to a trial of surgery alone vs. surgery with post-operative radiation. The primary endpoint is a second surgery to the same site within 12 months. Secondary outcomes include quality of life, pain and functional outcome markers, radiation or re-irradiation as applicable, a second surgery within 24 months for those patients alive, overall survival and cost effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Is the patient 18 years of age or older at the time of randomization?
* Does the patient have histologically or cytologically proven malignancy?
* Does the patient have imaging confirming presence of bone metastases corresponding to clinically painful area?
* Does the patient have established bone metastatic pathological fracture(s) lower extremity OR has impending pathological fracture(s)?
* Does patient have KPS ≥40 with estimated survival of ≥ 6 months?
* Was informed consent obtained?

Exclusion Criteria:

* Did the patient have a prior impending or prior pathological fracture to the site and was previously fixed with orthopaedic surgery?
* Did the patient receive prior radiation to the site (external beam or stereotactic body radiation)?
* Did the patient have a radio-resistant tumor (renal cell carcinoma or melanoma)?
* Did the patient plan for radical resection of the bone metastases?
* Did the patient receive or is planning to receive other intra-operative tumor ablative therapies?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Subsequent surgery after primary surgery | 12 months following the date of primary surgery
  Requirement of a subsequent surgery

SECONDARY OUTCOMES:
Re-irradiation/radiation | Weeks 2 & 6, Months 3, 6, 12, 18, and 24
  Requirement for re-irradiation in arm 2 or radiation in arm 1
Subsequent surgery (between 13 months and 24 months) | Between 13 months and 24 months following date of primary surgery
  Requirement of subsequent surgery past 12 months (between 13 months and 24 months)
Post-operative functional status and Karnofsky Performance Status (KPS) | Weeks 2 & 6, Months 3, 6, 12, 18, and 24
  The best, median, and worst post-operative functional status and KPS will be derived for each patient, and the Wilcoxin rank sum test will be used to compare the difference between treatment arms
Post-operative pain and analgesic use | Weeks 2 & 6, Months 3, 6, 12, 18, and 24
  The lowest, median, and worst post-operative pain score will be derived for each patient, and the Wilcoxin rank sum test will be used to compare the difference between treatment arms. The cumulative and mean of analgesic use will presented by treatment arm.
Radiologically determined local progression | Months 3, 6, 12, 18, and 24
  Time to radiological local disease progression is defined as the time from randomization to the date of documented radiological logical disease progression or death whichever comes first.
Quality of life through functional ability | Day of randomization, weeks 2 and 6, months 3, 6, 12, 18, and 24
  Quality of life measured measured using EORTC quality of life questionnaire (QLQ)-C15-Pal and EORTC quality of life questionnaire (QLQ)-BM22. This questionnaire includes for multi-item scales and six individual items. All items were scaled from 1 (not at all) to 4 (very much) in which a higher score indicates greater distress in symptom scales while a higher score in functional scale indicates greater functional ability. The EORTC QLQ-BM22 is a 22-item module that addresses disease symptoms related to bone metastasis. It has four subscales (painful sites, pain characteristics, functional interference and psychosocial aspects). All items were scaled from 1 (not at all) to 4 (very much), in which a higher score indicates greater distress in symptom scales while a higher score in functional scale indicates greater functional ability
Overall survival | Weeks 2 & 6, Months 3, 6, 12, 18, and 24
  Overall survival is defined as the time from randomization to the date of death from any cause, or censored at their last known alive data before or on data cutoff date
Cost-effectiveness | Weeks 2 & 6, Months 3, 6, 12, 18, and 24
  Determination of the incremental cost-effectiveness by prospectively collecting economic and resource utilization information. The objective is to determine an incremental cost effectiveness ratio reported as a cost per subsequent surgery avoided for both treatment arms. The mean overall cost per patient for each of the two study treatment arms will be calculated to determine the addition cost per surgery avoided.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Henry, MD FRCS(C), Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided